CLINICAL TRIAL: NCT06648460
Title: Multimodal Differences in Effort-based Decision-Making in Depression - - Brain Behavior Quantification and Synchronization
Brief Title: Multimodal Differences in Effort-based Decision-Making in Depression
Acronym: BBQS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Emory University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H24306
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Depression; Anhedonia
Keywords: Effort-based decision-making; Physical Effort
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: This is a single group study in which individuals with depression and matched controls will perform an effort-based decision-making task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effort-based decision-making (Other): Participants perform a virtual-reality-based task in which they expend effort to receive virtual rewards.
  Interventions: Other: Effort-based Decision-Making Task

INTERVENTIONS:
Other: Effort-based Decision-Making Task — Virtual Reality-based multi-stage task in which individuals must explore distinct "rooms" in a virtual environment that vary in the amount of effort (walking) and reward (points) they receive.

SUMMARY:
Major depressive disorder (MDD) is a serious condition that causes long-term symptoms such as feeling sad, losing interest in activities, and having thoughts of self-harm. Difficulty in making an effort is a key factor in functional impairment. Current methods to evaluate this difficulty use clinical assessments and computer-based tasks, but there is a gap between the measurements and real-life behavior. To address this, the study team proposes creating an instrumented behavioral test, HORMES, to objectively assess reduced motivation during everyday activities and measure physiological responses. The study will examine differences in brain activity, autonomic system function, and metabolic energy expenditure in patients with major depression during a decision-making task that involves physical effort.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a debilitating neuropsychiatric condition characterized by multiple chronic symptoms, including sad mood, anhedonia, psychomotor symptoms, and suicidal thoughts. MDD induces significant personal and societal suffering, becoming the largest contributor to the overall disease burden in developed countries. There is clearly an urgent need to advance our understanding of MDD and its constituent symptoms. Of these, the inability to expend effort have proven harder to treat than mood-related symptoms and are key predictors of functional impairment and disease burden. The biological mechanisms that contribute to this impairment are not fully understood. Addressing this gap in knowledge will be helpful in developing therapy, including novel brain stimulation therapies that offer the ability to target brain circuits precisely.

Current evaluation approaches to characterizing reduced motivation rely on clinical assessments of patient symptoms through interviews and observation. While these typically assess functions relevant to patient quality of life, these assessments may be confounded by biases. On the other hand, translational research focuses on characterizing symptoms using computer-based tasks that provide quantitative objective markers (e.g., reaction time in pressing a key on a keyboard) but may not reflect real-life situations. In addition, studies investigating brain mechanisms often use functional magnetic resonance imaging (fMRI), which requires patients to be stationary. Thus, there is a fundamental disconnect between measurements of behavior and the behavior itself under study.

To overcome these limitations, the study team envisions developing an instrumented behavioral assay, HORMES, that allows the objective assessment of reduced motivation during naturalistic behavior with concurrent measurements of the central and autonomic nervous systems as well as metabolic energy expenditure. This assay will utilize a CAREN system at Human Augmentation Core, a core facility available at Georgia Tech that is currently used for biomechanics research.

The proposed study will investigate differences in brain activity, autonomic system function, and metabolic energy expenditure in patients with major depression and matched controls during an effort-based decision-making task. The study team will collect multiple physiological measures - brain activity, cardiac activity, breathing activity, and energy expenditure in patients with major depression when they walk on a treadmill. Biomechanical information will be obtained using motion capture. The amount of effort they will need to expend will be varied by adjusting the treadmill's incline. These measures will be compared against those from a control group with age, gender, and BMI-matched healthy individuals.

The outcome of this study will inform what differences exist between healthy individuals and individuals with depression. The participants will be recruited from the Atlanta metro area and will all be allocated to the intervention. which is a behavioral task. The task requires participants to maximize rewards by choosing to pursue actions of different levels of physical effort (walking).

ELIGIBILITY:
Inclusion Criteria:

* Matched control group

  * 18-65 years old
  * Able-bodied
  * Fluent in English
  * Able to give written and verbal informed consent to the proposed experiment
  * Able to comprehend the study procedure, potential risks, and benefits
* Group with depression

  * Diagnosed with major depression
  * Quick Inventory of Depression Symptomology (QIDS) score > 5
  * 18-65 years old
  * Able-bodied
  * Fluent in English
  * Able to give written and verbal informed consent to the proposed experiment
  * Able to comprehend the study procedure, potential risks, and benefits

Exclusion Criteria:

* Matched control group

  * Current diagnosed psychiatric disorder (e.g., anxiety, depression, bipolar disorder)
  * Current pregnancy
  * BMI > 35
  * Currently on antipsychotics
* Group with depression

  * Diagnosed with psychotic symptoms
  * Diagnosed with other neurological or psychiatric disorders
  * Current pregnancy
  * BMI > 35
  * Currently on antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Time spent in high-effort "rooms" | 1 day
  Participants will be measured on how much time they spend in "rooms" that require high effort in the form of walking on an inclined treadmill as a proportion of the total duration of the task. This measures the willingness of participants to engage in effortful behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Rozell, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Georgia Tech Manufacturing Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in the NIMH Data Archive (NDA) at the end of the project. De-identified data sets will be anonymized prior to posting on the public repository. Shared data will include behavioral task outcomes, physiological data, and participant demographics.